CLINICAL TRIAL: NCT03165994
Title: A Phase 2 Study of APX005M in Combination With Concurrent Chemoradiation as Neoadjuvant Therapy for Resectable Esophageal and Gastroesophageal Junction Cancers
Brief Title: APX005M With Concurrent Chemoradiation for Resectable Esophageal and Gastroesophageal Junction Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apexigen America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX005M-006
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer; GastroEsophageal Cancer
Keywords: esophagus; gastroesophageal junction; T1-3N0-1; GE junction
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sotigalimab; Radiotherapy; Paclitaxel; Carboplatin; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Non-comparative, open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APX005M With Standard of Care Chemoradiation (Experimental): Participants will receive standard of care chemoradiation, consisting of:
  * External beam radiation in daily fractions (28 fractions) from Weeks 1-6, administered once per day up to 5 days/week.
  * Carboplatin (area under the carboplatin plasma concentration versus time curve = 2) and paclitaxel (50 mg/m^2) chemotherapy intravenously (IV) over 1 hour, once weekly, from Weeks 1-5.
  The participants also will receive concurrent 0.3 mg/kg APX005M IV over 1 hour, once weekly, on Weeks 1, 2, 4, and 6 (2-3 days after chemoradiation).
  Surgical resection of the tumor will be planned from Week 10 up to approximately Week 17, as indicated in the protocol amendment under which each participant is enrolled.
  Interventions: Drug: APX005M; Radiation: Radiation Therapy; Drug: Paclitaxel; Drug: Carboplatin; Procedure: Surgical resection of tumor

INTERVENTIONS:
Drug: APX005M — APX005M IV infusion
  Other Names: CD40 Agonistic Monoclonal Antibody; PYX-107; Sotigalimab
Radiation: Radiation Therapy — Radiation therapy, total dose 5040cGy in 180cGy fractions
  Other Names: Radiotherapy
Drug: Paclitaxel — Paclitaxel IV infusion
  Other Names: Taxol
Drug: Carboplatin — Carboplatin IV infusion
  Other Names: Paraplatin
Procedure: Surgical resection of tumor — Surgical removal of the tumor will occur between weeks 10-17
  Other Names: Surgery; Operation

SUMMARY:
This pilot phase II trial studies the therapeutic effects and side effects of CD40 agonistic monoclonal antibody APX005M when combined with chemotherapy and radiation therapy, and to see how well they work to reduce or remove esophageal or gastroesophageal (GE) cancers when given before surgery in treating patients with esophageal cancer or GE cancer than can be removed by surgery. APX005M is intended to stimulate the body's own immune system so that the immune cells can more effectively invade and destroy the tumor, adding to the benefits of the chemotherapy and radiation therapy. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving APX005M, chemotherapy, and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
Primary Objective:

To assess the efficacy of this novel combination, as measured by the pathologic complete response (pCR) rate.

Secondary Objectives:

1. To further characterize the safety and feasibility of combining APX005M with SOC chemoradiation (external beam radiation in daily fractions, with concurrent weekly low-dose carboplatin/paclitaxel) in the neoadjuvant setting for patients with resectable esophageal and GE junction cancers.
2. To assess the efficacy of combining APX005M with SOC chemoradiation as measured by rates of R0 resection (microscopically negative margins, i.e., no tumor remains following surgery); and radiographic/metabolic response to neoadjuvant treatment on CT-PET.

Exploratory Objectives:

1. To identify possible predictive molecular or immune-based efficacy biomarkers for this novel combination.
2. To characterize and assess overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Histologically proven squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma of the esophagus or GE junction.
3. Surgically resectable (T1-3 Nx preferably by endoscopic ultrasound [EUS]). (Excluded: T1N0 tumors, cervical esophageal location, tumors invading the tracheobronchial tree or with fistula, distant disease that cannot be included in the radiation field or be resected at the time of esophagectomy).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. Adequate hematological, renal, and hepatic parameters.

Exclusion Criteria:

1. Any history of or current hematologic malignancy.
2. History of a second primary cancer is allowed in the event the cancer is curatively resected and there is no evidence of recurrence/metastatic disease x 1 year. Subjects who have a history of cervical or breast carcinoma in situ, localized prostate cancer, adequately treated basal cell or squamous cell carcinoma of the skin, or superficial bladder tumors [Ta, Tis & T1] are also allowed.
3. Major surgery within 4 weeks of first dose of investigational product.
4. Prior or concurrent treatment with any anticancer agent for the same cancer diagnosis.
5. Prior exposure to any immuno-oncology agents, including CD40/PD-1/PD-L1/CTLA-4 inhibitors (if any ambiguity, should be discussed with study principal investigator).
6. History of bone marrow transplantation.
7. History of autoimmune disorders with the exception of vitiligo or autoimmune thyroid disorders.
8. Chronic steroid dependency (prednisone equivalent > 10 mg/day). Any steroid use should be discontinued at least 2 weeks prior to initiation of study treatment.
9. Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months before first dose.
10. Known human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - MedStar Georgetown University Hospital (MGUH), Washington D.C., District of Columbia
  - New York University, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Renovatio Clinical, The Woodlands, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko AH, Chao J, Noel MS, Shankaran V, Sohal D, Crow M, Oberstein PE, Scott AJ, McRee AJ, Rocha Lima CMSP, Fong L, Keenan BP, Soto M, Filbert EL, Hsu FJ, Yang X. A Phase 2 Study of Sotigalimab, a CD40 Agonist Antibody, plus Concurrent Chemoradiation as Neoadjuvant Therapy for Esophageal and Gastroesophageal Junction Cancers. Cancer Res Commun. 2025 Feb 1;5(2):349-357. doi: 10.1158/2767-9764.CRC-24-0513. PMID 39907035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 participants were eligible for the study, of which 33 received treatment in the study, in the United States between October 2017 and February 2023.
Pre-assignment Details: The study consisted of:
  * Screening Period (within 28 days of Treatment Period Day 1).
  * Treatment Period (Weeks 1-6) sotigalimab with standard-of-care (SOC) chemoradiation (chemoRT) consisting of external beam radiation in daily fractions, with concurrent weekly low-dose carboplatin/paclitaxel.
  * Post-treatment Period inc. surgery (Weeks 7-17).
  * Post-operative Follow-up Period (Months 1, 3, and 6 post-operatively).
  * Overall Survival Follow-up Period (every 3 months for 18 months).
Groups:
- Sotigalimab With SOC ChemoRT: Participants received SOC chemoRT, consisting of:
  * External beam radiation in daily fractions (28 fractions) from Weeks 1-6, administered once per day up to 5 days/week.
  * Carboplatin (area under the carboplatin plasma concentration versus time curve [AUC] = 2) and paclitaxel (50 mg/m^2) chemotherapy intravenously (IV) over 1 hour, once weekly, from Weeks 1-5.
  The participants also received concurrent 0.3 mg/kg sotigalimab IV over 1 hour, once weekly, on Weeks 1, 2, 4, and 6 (2-3 days after chemoRT).
  Surgical resection of the tumor was planned to be performed from Week 10 up to approximately Week 17, as indicated in the protocol amendment under which each participant was enrolled.
Period: Overall Study
Arm/Group | Sotigalimab With SOC ChemoRT
Started | 33
Completed | 13
Not Completed | 20
Not completed — Confirmed Radiographic Disease Progression | 4
Not completed — Death | 2
Not completed — Non-Compliance With Study Treatment or Procedure Requirements | 3
Not completed — Physician Decision, other than adverse event (AE) | 9
Not completed — Participant or Legal Representative Withdraws Consent | 1
Not completed — Miscellaneous | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of sotigalimab and scheduled SOC of chemoradiation therapy.
Groups:
- Sotigalimab With SOC ChemoRT: Participants received SOC chemoRT, consisting of:
  * External beam radiation in daily fractions (28 fractions) from Weeks 1-6, administered once per day up to 5 days/week.
  * Carboplatin (AUC = 2) and paclitaxel (50 mg/m^2) chemotherapy IV over 1 hour, once weekly, from Weeks 1-5.
  The participants also received concurrent 0.3 mg/kg sotigalimab IV over 1 hour, once weekly, on Weeks 1, 2, 4, and 6 (2-3 days after chemoRT).
  Surgical resection of the tumor was planned to be performed from Week 10 up to approximately Week 17, as indicated in the protocol amendment under which each participant was enrolled.
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25
  Black or African | 1
  Asian | 5
  Other | 2
Tumor Histology [Count of Participants; unit: Participants]
  Squamous Cell Carcinoma | 8
  Adenocarcinoma | 25
Tumor Location [Count of Participants; unit: Participants] — Non-gastroesophageal (GE) Junction tumor location includes upper, middle, and lower thirds of the esophagus.
  Participants
    GE Junction | 15
    Non-GE Junction | 18

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR) Rate (%) Overall
Description: The pCR was defined as post-neoadjuvant pathologic tumour, node, metastasis (ypTNM) (after chemoRT; after surgery) with T0, N0 stages. pCR rate was defined as the percentage of participants who achieved a pCR at surgery, as assessed by the Investigator.
  * T0: No evidence of primary tumor.
  * N0: Cancer has not spread to nearby lymph nodes.
  An exact Clopper-Pearson lower 95% confidence limit was used to test the null hypothesis that the pCR rate is ≤30%.
Time Frame: At time of surgery, up to a maximum of 261 days
Population: Efficacy Population: All participants who were eligible, received neoadjuvant sotigalimab and chemoRT followed by surgery, or had their planned surgery aborted due to the discovery of progressive disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
percentage of participants | 37.9 [20.7 to 57.7]

2. Primary Outcome: pCR Rate (%) by Baseline Histologic Subgroup
Description: The pCR was defined as ypTNM (after chemoRT; after surgery) with T0, N0 stages. pCR rate was defined as the percentage of participants who achieved a pCR at surgery, as assessed by the Investigator.
  An exact Clopper-Pearson lower 95% confidence limit was used to test the null hypothesis that the pCR rate is ≤30%.
Time Frame: At time of surgery, up to a maximum of 261 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
percentage of participants
  Squamous Cell Carcinoma: number analyzed (Participants) | 5
  Squamous Cell Carcinoma | 60.0 [14.7 to 94.7]
  Adenocarcinoma: number analyzed (Participants) | 24
  Adenocarcinoma | 33.3 [15.6 to 55.3]

3. Primary Outcome: pCR Rate (%) by Baseline Tumor Location Subgroup
Description: as for outcome 2
Time Frame: At time of surgery, up to a maximum of 261 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
percentage of participants
  GE Junction: number analyzed (Participants) | 14
  GE Junction | 28.6 [8.4 to 58.1]
  Non-GE Junction: number analyzed (Participants) | 15
  Non-GE Junction | 46.7 [21.3 to 73.4]

4. Primary Outcome: pCR Rate (%) by Steroid Use Subgroup
Description: The pCR was defined as ypTNM (after chemoRT; after surgery) with T0, N0 stages. pCR rate was defined as the percentage of participants who achieved a pCR at surgery, as assessed by the Investigator. Steroids use: Yes was defined as participants with any steroid (ATC2 class corticosteroids for systemic use) from within 30 days of the first dose of sotigalimab to up to 7 days after the first dose and participants not fulfilling previous requirements are defined as Steroids use: No.
  An exact Clopper-Pearson lower 95% confidence limit was used to test the null hypothesis that the pCR rate is ≤30%.
Time Frame: At time of surgery, up to a maximum of 261 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
percentage of participants
  Steroid Use: Yes: number analyzed (Participants) | 16
  Steroid Use: Yes | 31.3 [11.0 to 58.7]
  Steroid Use: No: number analyzed (Participants) | 13
  Steroid Use: No | 46.2 [19.2 to 74.9]

5. Primary Outcome: pCR Rate (%) by Surgery Subgroup
Description: The pCR was defined as ypTNM (after chemoRT; after surgery) with T0, N0 stages. pCR rate was defined as the percentage of participants who achieved a pCR at surgery, as assessed by the Investigator.
  The subgroup of participants who had surgery before or at 16/17 weeks were defined as start of study treatment to surgery date from the surgical resection form, less than or equal to 17 weeks (119 days = 17 weeks * 7 days) or participants who were scheduled to have surgery but had their procedure aborted due to progressive disease at the time of the procedure or immediately before and did not have surgery because of metastasis. The subgroup of participants who had surgery after Week 17 were defined as start of study treatment to surgery date from the surgical resection form, greater than 17 weeks.
  An exact Clopper-Pearson lower 95% confidence limit was used to test the null hypothesis that the pCR rate is ≤30%.
Time Frame: At time of surgery, up to a maximum of 261 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
percentage of participants
  Surgery Before or at Week 16-17: number analyzed (Participants) | 21
  Surgery Before or at Week 16-17 | 28.6 [11.3 to 52.2]
  Surgery After Week 17: number analyzed (Participants) | 8
  Surgery After Week 17 | 62.5 [24.5 to 91.5]

6. Secondary Outcome: Rate (%) of R0 Resection Overall
Description: R0 was defined as the absence of gross and microscopic tumor involvement in the surgical margins i.e., no tumor remains following surgery. Rate of R0 resection was defined as the percentage of participants who achieved R0 following surgical resection.
Time Frame: At time of surgery, up to a maximum of 261 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
percentage of participants | 86.2

7. Secondary Outcome: Rate (%) of R0 Resection by Baseline Histologic Subgroup
Description: as for outcome 6
Time Frame: At time of surgery, up to a maximum of 261 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
percentage of participants
  Squamous Cell Carcinoma: number analyzed (Participants) | 5
  Squamous Cell Carcinoma | 100
  Adenocarcinoma: number analyzed (Participants) | 24
  Adenocarcinoma | 83.3

8. Secondary Outcome: Pathologic Stage at Time of Surgery
Description: Pathologic staging was assessed via ypTNM (after chemoRT and surgery):
  * Tumor Stage (TX, T0, T1, T1a, T1b, T2, T3, T4, T4a, T4b) refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it had grown into the wall of the esophagus.
  * Node Stage (NX, N0, N1, N2, N3) refers to the number and location of lymph nodes that cancer has spread to. The higher the number after the N, the more lymph nodes that contained cancer cells.
  * Metastasis Stage (M0, M1) refers to whether the cancer had not spread (M0) or spread (M1) to other parts of the body.
  * Stage group (0, I, IA, IB, II, IIA, IIB, III, IIIA, IIIB, IV, IVA, IVB) are based on the TNM stages detailed above. The higher the number, the more advanced the cancer was.
  For each category, a lower stage/group represents a better outcome.
Time Frame: At time of surgery, up to a maximum of 261 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
Participants
  Tumor Stage: Missing | 2
  Tumor Stage: T0 | 12
  Tumor Stage: T1a | 1
  Tumor Stage: T2 | 5
  Tumor Stage: T3 | 9
  Node Stage: Missing | 2
  Node Stage: N0 | 21
  Node Stage: N1 | 3
  Node Stage: N2 | 2
  Node Stage: N3 | 1
  Metastasis Stage: Missing | 2
  Metastasis Stage: M0 | 27
  Stage Group: Missing | 13
  Stage Group: I | 2
  Stage Group: IA | 1
  Stage Group: II | 6
  Stage Group: III | 1
  Stage Group: IIIA | 2
  Stage Group: IIIB | 3
  Stage Group: IVA | 1

9. Secondary Outcome: Radiographic/Metabolic Response to Neoadjuvant Treatment on Computed Tomography (CT)/CT-Positron Emission Tomography (PET) (CT-PET) Overall
Description: Response was adjudicated by the investigator; based on combination of change in wall thickening; size of regional lymph nodes; and metabolic activity of involved areas.
  As the population does not typically have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST), radiographic/metabolic response was described in qualitative terms (responding/ stable, unchanged/ progressing/ not evaluable).
Time Frame: At time of surgery, up to a maximum of 261 days, 3 and 6 months post-operatively, and End of Study Visit (maximum of 6 months post-operatively)
Population: Efficacy Population: All participants who were eligible, received neoadjuvant sotigalimab and chemoRT followed by surgery, or had their planned surgery aborted due to the discovery of progressive disease. Participants with data available at each time point are presented. Participants included at End of Study Visit discontinued prior to completion of Postoperative Follow-up/Month 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
Participants
  At Time of Surgery: Missing | 0
  At Time of Surgery: Responding | 22
  At Time of Surgery: Stable/Unchanged | 5
  At Time of Surgery: Progressing | 1
  At Time of Surgery: Not Evaluable | 1
  Postoperative Follow-up/Month 3: number analyzed (Participants) | 18
  Postoperative Follow-up/Month 3: Missing | 3
  Postoperative Follow-up/Month 3: Responding | 9
  Postoperative Follow-up/Month 3: Stable/Unchanged | 2
  Postoperative Follow-up/Month 3: Progressing | 1
  Postoperative Follow-up/Month 3: Not Evaluable | 3
  Postoperative Follow-up/Month 6: number analyzed (Participants) | 13
  Postoperative Follow-up/Month 6: Missing | 3
  Postoperative Follow-up/Month 6: Responding | 6
  Postoperative Follow-up/Month 6: Stable/Unchanged | 1
  Postoperative Follow-up/Month 6: Progressing | 2
  Postoperative Follow-up/Month 6: Not Evaluable | 1
  End of Study Visit: number analyzed (Participants) | 9
  End of Study Visit: Missing | 2
  End of Study Visit: Responding | 2
  End of Study Visit: Stable/Unchanged | 0
  End of Study Visit: Progressing | 3
  End of Study Visit: Not Evaluable | 2

10. Secondary Outcome: Radiographic/Metabolic Response to Neoadjuvant Treatment on CT-PET by Baseline Histologic Subgroup
Description: Response was adjudicated by the investigator; based on combination of change in wall thickening; size of regional lymph nodes; and metabolic activity of involved areas.
  As the population does not typically have measurable disease by RECIST, radiographic/metabolic response was described in qualitative terms (responding/ stable, unchanged/ progressing/ not evaluable).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
Participants
  Squamous Cell Carcinoma: At Time of Surgery: number analyzed (Participants) | 5
  Squamous Cell Carcinoma: At Time of Surgery: Missing | 0
  Squamous Cell Carcinoma: At Time of Surgery: Responding | 5
  Squamous Cell Carcinoma: At Time of Surgery: Stable/Unchanged | 0
  Squamous Cell Carcinoma: At Time of Surgery: Progressing | 0
  Squamous Cell Carcinoma: At Time of Surgery: Not Evaluable | 0
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 3: number analyzed (Participants) | 3
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 3: Missing | 1
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 3: Responding | 1
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 3: Stable/Unchanged | 0
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 3: Progressing | 0
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 3: Not Evaluable | 1
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 6: number analyzed (Participants) | 3
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 6: Missing | 0
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 6: Responding | 1
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 6: Stable/Unchanged | 0
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 6: Progressing | 1
  Squamous Cell Carcinoma: Postoperative Follow-up/Month 6: Not Evaluable | 1
  Squamous Cell Carcinoma: End of Study Visit: number analyzed (Participants) | 1
  Squamous Cell Carcinoma: End of Study Visit: Missing | 0
  Squamous Cell Carcinoma: End of Study Visit: Responding | 0
  Squamous Cell Carcinoma: End of Study Visit: Stable/Unchanged | 0
  Squamous Cell Carcinoma: End of Study Visit: Progressing | 1
  Squamous Cell Carcinoma: End of Study Visit: Not Evaluable | 0
  Adenocarcinoma: At Time of Surgery: number analyzed (Participants) | 24
  Adenocarcinoma: At Time of Surgery: Missing | 0
  Adenocarcinoma: At Time of Surgery: Responding | 17
  Adenocarcinoma: At Time of Surgery: Stable/Unchanged | 5
  Adenocarcinoma: At Time of Surgery: Progressing | 1
  Adenocarcinoma: At Time of Surgery: Not Evaluable | 1
  Adenocarcinoma: Postoperative Follow-up/Month 3: number analyzed (Participants) | 15
  Adenocarcinoma: Postoperative Follow-up/Month 3: Missing | 2
  Adenocarcinoma: Postoperative Follow-up/Month 3: Responding | 8
  Adenocarcinoma: Postoperative Follow-up/Month 3: Stable/Unchanged | 2
  Adenocarcinoma: Postoperative Follow-up/Month 3: Progressing | 1
  Adenocarcinoma: Postoperative Follow-up/Month 3: Not Evaluable | 2
  Adenocarcinoma: Postoperative Follow-up/Month 6: number analyzed (Participants) | 10
  Adenocarcinoma: Postoperative Follow-up/Month 6: Missing | 3
  Adenocarcinoma: Postoperative Follow-up/Month 6: Responding | 5
  Adenocarcinoma: Postoperative Follow-up/Month 6: Stable/Unchanged | 1
  Adenocarcinoma: Postoperative Follow-up/Month 6: Progressing | 1
  Adenocarcinoma: Postoperative Follow-up/Month 6: Not Evaluable | 0
  Adenocarcinoma: End of Study Visit: number analyzed (Participants) | 8
  Adenocarcinoma: End of Study Visit: Missing | 2
  Adenocarcinoma: End of Study Visit: Responding | 2
  Adenocarcinoma: End of Study Visit: Stable/Unchanged | 0
  Adenocarcinoma: End of Study Visit: Progressing | 2
  Adenocarcinoma: End of Study Visit: Not Evaluable | 2

11. Secondary Outcome: Radiographic/Metabolic Response to Neoadjuvant Treatment on CT-PET by Baseline Tumor Location Subgroup
Description: as for outcome 10
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 29
Participants
  GE Junction: At Time of Surgery: number analyzed (Participants) | 14
  GE Junction: At Time of Surgery: Missing | 0
  GE Junction: At Time of Surgery: Responding | 10
  GE Junction: At Time of Surgery: Stable/Unchanged | 3
  GE Junction: At Time of Surgery: Progressing | 1
  GE Junction: At Time of Surgery: Not Evaluable | 0
  GE Junction: Postoperative Follow-up/Month 3: number analyzed (Participants) | 9
  GE Junction: Postoperative Follow-up/Month 3: Missing | 2
  GE Junction: Postoperative Follow-up/Month 3: Responding | 4
  GE Junction: Postoperative Follow-up/Month 3: Stable/Unchanged | 1
  GE Junction: Postoperative Follow-up/Month 3: Progressing | 0
  GE Junction: Postoperative Follow-up/Month 3: Not Evaluable | 2
  GE Junction: Postoperative Follow-up/Month 6: number analyzed (Participants) | 5
  GE Junction: Postoperative Follow-up/Month 6: Missing | 2
  GE Junction: Postoperative Follow-up/Month 6: Responding | 1
  GE Junction: Postoperative Follow-up/Month 6: Stable/Unchanged | 1
  GE Junction: Postoperative Follow-up/Month 6: Progressing | 1
  GE Junction: Postoperative Follow-up/Month 6: Not Evaluable | 0
  GE Junction: End of Study Visit: number analyzed (Participants) | 5
  GE Junction: End of Study Visit: Missing | 1
  GE Junction: End of Study Visit: Responding | 1
  GE Junction: End of Study Visit: Stable/Unchanged | 0
  GE Junction: End of Study Visit: Progressing | 3
  GE Junction: End of Study Visit: Not Evaluable | 0
  Non-GE Junction: At Time of Surgery: number analyzed (Participants) | 15
  Non-GE Junction: At Time of Surgery: Missing | 0
  Non-GE Junction: At Time of Surgery: Responding | 12
  Non-GE Junction: At Time of Surgery: Stable/Unchanged | 2
  Non-GE Junction: At Time of Surgery: Progressing | 0
  Non-GE Junction: At Time of Surgery: Not Evaluable | 1
  Non-GE Junction: Postoperative Follow-up/Month 3: number analyzed (Participants) | 9
  Non-GE Junction: Postoperative Follow-up/Month 3: Missing | 1
  Non-GE Junction: Postoperative Follow-up/Month 3: Responding | 5
  Non-GE Junction: Postoperative Follow-up/Month 3: Stable/Unchanged | 1
  Non-GE Junction: Postoperative Follow-up/Month 3: Progressing | 1
  Non-GE Junction: Postoperative Follow-up/Month 3: Not Evaluable | 1
  Non-GE Junction: Postoperative Follow-up/Month 6: number analyzed (Participants) | 8
  Non-GE Junction: Postoperative Follow-up/Month 6: Missing | 1
  Non-GE Junction: Postoperative Follow-up/Month 6: Responding | 5
  Non-GE Junction: Postoperative Follow-up/Month 6: Stable/Unchanged | 0
  Non-GE Junction: Postoperative Follow-up/Month 6: Progressing | 1
  Non-GE Junction: Postoperative Follow-up/Month 6: Not Evaluable | 1
  Non-GE Junction: End of Study Visit: number analyzed (Participants) | 4
  Non-GE Junction: End of Study Visit: Missing | 1
  Non-GE Junction: End of Study Visit: Responding | 1
  Non-GE Junction: End of Study Visit: Stable/Unchanged | 0
  Non-GE Junction: End of Study Visit: Progressing | 0
  Non-GE Junction: End of Study Visit: Not Evaluable | 2

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events which started on or after the first infusion of study treatment (Carboplatin/Paclitaxel/Sotigalimab/Radiotherapy) until 100 days after receiving the last dose of study treatment, death, or initiation of new anticancer therapy, whichever occurs first. Laboratory values that were considered clinically significant were reported as adverse events.
Time Frame: Up to approximately 20 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Sotigalimab With SOC ChemoRT
Number analyzed (Participants) | 33
Participants | 33

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrollment to completion of the overall survival follow-up period; approximately 28 months. Adverse events were collected from the first infusion of study treatment until 100 days after receiving the last dose of study treatment, death, or initiation of new anticancer therapy, whichever occurs first; up to approximately 20 weeks.
Description: All-cause mortality was collected for all participants enrolled/randomized in the study. Adverse events were collected for all participants in the Safety Population who received at least one dose of sotigalimab and scheduled SOC of chemoradiation therapy. Adverse events are presented regardless of causal relationship to any of the study treatments.
Arm/Group | Sotigalimab With SOC ChemoRT
All-Cause Mortality (participants affected / at risk) | 7/33
Serious Adverse Events (participants affected / at risk) | 16/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotigalimab With SOC ChemoRT (N=33)
Nausea (Gastrointestinal disorders) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 3 (3)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Impaired healing (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotigalimab With SOC ChemoRT (N=33)
Nausea (Gastrointestinal disorders) | 23 (40)
Constipation (Gastrointestinal disorders) | 16 (20)
Diarrhoea (Gastrointestinal disorders) | 15 (21)
Vomiting (Gastrointestinal disorders) | 13 (28)
Dysphagia (Gastrointestinal disorders) | 11 (12)
Oesophagitis (Gastrointestinal disorders) | 9 (9)
Oesophageal pain (Gastrointestinal disorders) | 7 (8)
Odynophagia (Gastrointestinal disorders) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Haematochezia (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 24 (41)
Chills (General disorders) | 16 (31)
Pyrexia (General disorders) | 8 (13)
Chest discomfort (General disorders) | 2 (2)
Influenza like illness (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 15 (29)
Leukopenia (Blood and lymphatic system disorders) | 14 (39)
Neutropenia (Blood and lymphatic system disorders) | 14 (35)
Anaemia (Blood and lymphatic system disorders) | 9 (17)
Lymphopenia (Blood and lymphatic system disorders) | 5 (17)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 14 (26)
Alanine aminotransferase increased (Investigations) | 14 (23)
Blood alkaline phosphatase increased (Investigations) | 6 (9)
Weight decreased (Investigations) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (17)
Dehydration (Metabolism and nutrition disorders) | 8 (9)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Headache (Nervous system disorders) | 7 (11)
Dizziness (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (13)
Radiation skin injury (Injury, poisoning and procedural complications) | 2 (2)
Hypotension (Vascular disorders) | 7 (8)
Flushing (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Cytokine release syndrome (Immune system disorders) | 8 (12)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT03165994/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03165994/SAP_001.pdf